CLINICAL TRIAL: NCT00743444
Title: A Double-blind, Placebo Controlled, Randomized, Two Centre Phase IIA Pharmacodynamic Cross-over Study to Assess the Effect of AZD3355, 65 mg Bid, on Transient Lower Esophageal Sphincter Relaxations (TLESRs) in GERD Patients With an Incomplete Response to PPI Treatment
Brief Title: TLESR-impedance Study in Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: D9120C00020
Record Dates: First submitted 2008-08-26; First posted 2008-08-28 (Estimated); Results first posted 2011-06-10 (Estimated); Last update posted 2013-07-22 (Estimated); Status verified 2013-07

CONDITIONS: Reflux Episodes
Keywords: GERD; transient lower esophageal sphincter relaxations (TLESRs); reflux
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — lesogaberan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): AZD3355
  Interventions: Drug: AZD3355
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD3355 — 65 mg capsules, oral, 3 single doses
  Other Names: Lesogaberan
  Arms: 1
Drug: Placebo — capsules, oral, 3 single doses
  Arms: 2

SUMMARY:
The purpose of the study is to compare frequency and content of reflux episodes in patients with gastroesophageal reflux disease.

ELIGIBILITY:
Inclusion Criteria:

* Provision of written consent
* GERD patients, age 18-70 years, females must be postmenopausal or surgically sterilised
* 6 months history of GERD and incomplete response to PPI treatment

Exclusion Criteria:

* Insufficient symptom burden of the reflux disease evaluated by questionnaires
* S-creatinine >1.2 times upper limit of normal
* History of heart disease
* Prior surgery of the upper GI tract

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2007-02; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eva Ersdal, PhD, Study Director — AstraZeneca R&D, Mölndal, Sweden; Daniel Sifrim, MD, PhD, Principal Investigator — Center for Gastroenterological Research, Belgium

REFERENCES:
- [Derived] Boeckxstaens GE, Beaumont H, Mertens V, Denison H, Ruth M, Adler J, Silberg DG, Sifrim D. Effects of lesogaberan on reflux and lower esophageal sphincter function in patients with gastroesophageal reflux disease. Gastroenterology. 2010 Aug;139(2):409-17. doi: 10.1053/j.gastro.2010.04.051. Epub 2010 May 5. PMID 20451523

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 42 patients in 2 countries were enrolled in the study. 27 patients were randomised to treatment. 2 patients discontinued prematurely, 1 due to low Lower Esophageal Sphincter Pressure (LESP)/catheter placement problems, and 1 due to nausea/vomiting. Thus, 25 patients completed the study, 10 in Belgium and 15 in the Netherlands.
Groups:
- AZD3355 First, Then Placebo; Placebo First, Then AZD3355: 65 mg drug or placebo capsules, oral, 3 single doses
Period: First Intervention
Arm/Group | AZD3355 First, Then Placebo | Placebo First, Then AZD3355
Started | 14 | 13
Completed | 14 | 12
Not Completed | 0 | 1
Not completed — Catheter placement problems | 0 | 1
Period: Washout Period
Arm/Group | AZD3355 First, Then Placebo | Placebo First, Then AZD3355
Started | 14 | 12
Completed | 14 | 11
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1
Period: Second Intervention
Arm/Group | AZD3355 First, Then Placebo | Placebo First, Then AZD3355
Started | 14 | 11
Completed | 14 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Entire Study Population: Includes groups randomized to received Drug first and Placebo first.
Arm/Group | Entire Study Population
Number analyzed (Participants) | 27
Age Continuous [Mean (Standard Deviation); unit: years] | 51.6 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 16

OUTCOME MEASURES:

1. Primary Outcome: Number of Transient Lower Esophageal Sphincter Relaxations (TLESRs) 0-3 Hours Post Meal, Post Third Dose
Description: The number of relaxations for each patient in each period was determined from manometric tracings according to previously published criteria (R.H. Holloway, R. Penagini and A.C. Ireland, Criteria for objective definition of transient lower esophageal sphincter relaxation, Am J Physiol 268 (1995), pp. G128-G133).
  The analysis of the number of TLESRs was based on an analysis of variance (ANOVA) for log-transformed data. The 95% level confidence interval (CI) limits were transformed back to the original scale to give CIs for the geometric mean for each treatment.
Time Frame: 0-3 hours post meal, post third dose
Population: Per Protocol Analysis Set (PP). From the safety analysis set with 27 patients, the PP excludes 2 patients since they discontinued prematurely from the study. Additionally, 4 patients were excluded from the primary analysis; 1 due to catheter placement problems, 1 due to error in dose administration, 1 due to low LESP, 1 due to multiple swallowing.
Measure: Geometric Mean (95% Confidence Interval); unit: Relaxations
Groups:
- AZD3355: 65 mg drug capsules, oral, 3 single doses
- Placebo: placebo capsules, oral, 3 single doses
Arm/Group | AZD3355 | Placebo
Number analyzed (Participants) | 21 | 21
Relaxations | 11.6 [9.40 to 14.3] | 15.5 [12.6 to 19.1]

2. Secondary Outcome: Total Number Reflux Episodes 0-24 Hours Post First Dose
Description: Number of reflux episodes assessed during the 24-hour ambulatory impedance-pH recording.
Time Frame: 0-24 hours
Population: Per Protocol Analysis Set (PP). From the safety analysis set with 27 patients, the PP excludes 2 patients since they discontinued prematurely from the study. Additionally, 4 patients were excluded from this analysis; 1 due to catheter placement problems, 1 due to error in dose administration, 2 due to insufficient impedance/pH recording time.
Measure: Geometric Mean (95% Confidence Interval); unit: Episodes
Arm/Group | AZD3355 | Placebo
Number analyzed (Participants) | 21 | 21
Episodes | 30.6 [20.9 to 44.9] | 50.5 [34.5 to 74.1]

3. Secondary Outcome: Area Under the Plasma Concentration vs. Time Curve (AUCtau) During 0-12 Hours Post First Dose Calculated by the Log/Linear Trapezoidal Method.
Description: The AUCtau was calculated for each patient in the period with AZD3355 treatment by the Log-Linear Trapezoidal Method. The descriptive geometric mean of the individual AUCtau values is reported here.
Time Frame: 0-12 hours post first dose
Population: Per Protocol Analysis Set (PP). From the safety analysis set with 27 patients, the PP excludes 2 patients since they discontinued prematurely from the study. Additionally, 1 patient was excluded from the pharmacokinetic analysis due to error in dose administration at dose 2.
Measure: Geometric Mean (Standard Deviation); unit: μmol*hours / L
Arm/Group | AZD3355
Number analyzed (Participants) | 24
μmol*hours / L | 7.16 (2.36)

ADVERSE EVENTS:
Arm/Group | AZD3355 | Placebo
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/27
Other Adverse Events (participants affected / at risk) | 16/25 | 18/27
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AZD3355 (N=25) | Placebo (N=27)
Abdominal Distension (Gastrointestinal disorders) | 3 | 1
Nausea (Gastrointestinal disorders) | 2 | 5
Nasopharyngitis (Infections and infestations) | 1 | 2
Dizziness (Nervous system disorders) | 3 | 1
Headache (Nervous system disorders) | 8 | 11
Paraesthesia (Nervous system disorders) | 5 | 3
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 2
Hot Flush (Vascular disorders) | 3 | 1
Flatulence (Gastrointestinal disorders) | 2 | 1
Feeling Hot (General disorders) | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
There is an agreement between PI and Sponsor (AZ) or its agents that restricts the PI's right to discuss/publish trial results after the trial is completed. The PI agrees to collaborate in good faith with AZ with regards to content and formation of any publication or disclosure to be made by PI and to pay due consideration to opinions offered by AZ.